CLINICAL TRIAL: NCT02027194
Title: Effects of Chinese Herbal Medicine for Treatment of Allergic Rhinitis: A Randomized Controlled Trial
Brief Title: Controlled Trial of Chinese Herbal Medicine to Treat Allergic Rhinitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Chien Wai-Tong, Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PhD thesis
Record Dates: First submitted 2014-01-02; First posted 2014-01-06 (Estimated); Last update posted 2015-03-13 (Estimated); Status verified 2015-03

CONDITIONS: Allergic Rhinitis
Keywords: Allergic Rhinitis; Chinese herbal medicine; Adolescents; Double-blinded; Randomized controlled trial
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cure-Allergic Rhinitis Syrup (Experimental): In syrup form, 20 ml once daily for 4 weeks
  Interventions: Drug: Cure-Allergic Rhinitis Syrup
- Yu-ping-fung San (Active Comparator): In syrup form, 20ml once daily for 4 weeks
  Interventions: Drug: Yu-ping-fung San
- Placebo group (Placebo Comparator): In syrup form (wheat powder with ginger and flavors), 20 ml once daily for 4 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cure-Allergic Rhinitis Syrup — Delivered one bottle for two weeks to the participants twice
  Other Names: CS group
  Arms: Cure-Allergic Rhinitis Syrup
Drug: Yu-ping-fung San — Delivered one bottle for 2-week usage to the participants twice
  Other Names: YS group
  Arms: Yu-ping-fung San
Drug: Placebo — Delivered one bottle (wheat power with favors) for 2-week usage to the participants twice
  Other Names: Placebo/Control
  Arms: Placebo group

SUMMARY:
The aim of this study is to test and compare the effectiveness between three groups - Cure-Allergic Rhinitis Syrup (CS), Yuk ping fung San (YS) and placebo groups - of adolescents (nursing students) with Allergic Rhinitis (AR) in improving their symptoms of AR, body constitution pattern and health-related quality of life.

• The hypothesis are to test the effectiveness of the CS treatment on these students' AR symptoms and quality of life at immediately, one month and two months after completion of the 4-week intervention, when compared with the YS treatment and placebo group.

1. Cure-Allergic Rhinitis Syrup (CS) group will show significantly reduction of AR symptoms over the 2-month follow-up, when compared to those in YS and placebo groups.
2. CS group will indicate a healthier body constitution pattern over the follow-up, when compared to those with YS and placebo group.
3. CS group will indicate significantly greater improvement of their quality of life over 2-month follow-up, when compared to those with YS and placebo group.

DETAILED DESCRIPTION:
Background

* Rhinitis (AR) is one of the most concerned public health problems worldwide, resulting from an inflammation of nasal membranes.
* Nursing students is one of the high risk groups, particularly when performing clinical practicum in hospitals in which they would contact with multiple allergens such as micro-organisms, detergents, chemical agents, and frequently used powdered latex gloves. More than 10% of these adolescents would present consistent AR symptoms such as nasal congestion, sneezing and sleep problems and In turn, these symptoms could affect their quality of life and academic performance.
* Non-compliance to medication or refusals to medical advice was common due to lack of efficacy, side effects, fear of being habit-forming, and/or expensive medical costs; and thus many preferred an alternative therapy for improved symptoms and bodily condition, and even full recovery.
* Chinese medicine treats the disease from the root, which is a complementary and alternative approach for holistic convalescence by changing unhealthy body constitution (health status) to healthy. However, little scientific evidence has been established for the treatment of AR with Chinese herbal medicine.
* This study aims to test the effects of two alternative treatments of Chinese herbal medicine, including Cure-Allergic Rhinitis Syrup (CS) and Yuk ping fung San, when compared with a placebo (i.e., wheat syrup with similar taste and smell) group, in reducing university nursing students' AR symptom severity and improving their quality of life and body constitution.

Methodology

* A double-blind randomized controlled trial with repeated-measures, three parallel groups design is adopted.
* Assessment and follow-ups would be taken place in an Integrative Health Clinic of The University under study.
* Stratified random sampling method in terms of the students' years of illness onset and gender has been used to allocate the subjects into one of the three study groups.
* Participants, assessor and researcher are concealed and blinded to the random group allocation, which would be performed by an independent clinic nurse.
* In order to maintain complete blinding, a clinic nurse will also administer the herbal medicine and keep the name list locked, and thus being confidential.
* Participants would be recruited from all of five full-time undergraduate nursing programs in School of Nursing of The University. After their eligibility for inclusion checked and baseline measurement performed with informed consent obtained, the participants would be grouped in terms of duration of the illness (0-2 years, 2-5 years and 5 or above years) and gender and then each would draw one labeled card from an opaque envelope (1=CS, 2=YS and 3=Placebo) from the clinic nurse to allocate them into one of the three groups.
* Quality of life and symptom severity would be measured with self-administered questionnaires, and body constitution assessment would be performed by an Traditional Chinese medicine (TCM) practitioner, at baseline and immediately, one-month and three-month after the 4-week intervention.

Sampling

* All full-time nursing students in The University under study who met the inclusion criteria and voluntary to participate in this study are the potential subjects.
* Sample size calculation has been calculated in the basis of similar Chinese herbal medicine effects in improving AR symptoms (primary outcome) in previous studies. Total sample size is 195 (n=65 per group) using G-Power based on the effect sizes (0.45) of two similar recent studies (Jung, 2011; Yang, 2010). Taking account of about 20% drop-outs, the estimated sample size becomes 234, thus 78 participants in each group.

Intervention

* Cure-Allergic Rhinitis Syrup (CS) and Yuk ping fung San (YS) are adopted as the two alternative treatments to be tested in this study, while the placebo group will be the controls in this study.
* Medication will be produced and provided by the researcher. CS contains 12 Chinese herbal medicines in one formula, combining 3 classical ancient formula of herbal medicine that are commonly used to enhance healthy body constitution. YS contains 6 herbal medicines, which are commonly used for AR treatment, while the placebo contains wheat powder, sugar and spicy taste of food (ginger).
* Boiling methods for CS and YS are the same, in which the herbal medicines will be boiled with 2000 ml of water for two hours after cleansing to about 500 ml herbal concoction.
* Participants would be asked to take 20 ml per dosage on each day, by diluting two spoons with a half cup of water either in the morning or at night, at their convenience.
* One bottle for two-week dosage would be offered after the first assessment at recruitment; and another bottle for the remaining 2-week dosage would be given during the first follow-up by the end of 2nd week (Interim assessment). Each participant would have to take in total of four weeks herbal medicine.

Ethical issues

* Ethical approval of this study will be obtained from the Human Subjects Research Ethics Sub-committee of The Hong Kong Polytechnic University.
* Written informed consent will be obtained from the respondents to show their willingness of participation. In order to enhance full understanding of the study before participation, an information sheet to describe in more details about the aim and procedure of the study will be given with explanations before signing the written consent.
* Study data and participant identity are kept anonymous and confidential. Data collected are limited in access by the researcher and clinic nurse for study purpose only. The data will be destroyed after completion of the study and thesis writing.
* Precaution of adverse effects would be taken on the herbal medicine selection (double-checked by an independent TCM practitioner), medicine formation (agreed by at least two TCM practitioners), time of boiling, and interim assessment (by one TCM practitioner) and weekly or bi-weekly face-to-face or telephone follow-ups (by the researcher). Students are reminded of reporting any discomfort and asking questions about the illness and the study. They are given the contact telephone of the researcher and would be referred to Western medicine or TCM practitioner for follow-up, as needed.
* All herbal medicine items should be within normal and recommended dosage. Any toxic effect of the herbal medicines used is reduced by long boiling and minimal dosage.
* Before random group allocation, all participants are assessed and confirmed with the body constitution pattern(s) by one TCM practitioner and history of allergy to herbal medicines, particularly those items adopted in the study, will be checked. Those with such allergies, inappropriate body constitution for the herbal medicines used, or very poor body condition, would be excluded.
* Monitoring of exceptional allergy such as skin rash and related discomforts would be performed over the first 2 weeks of syrup intake. At the end of the 1st and 3rd week of intervention, the researcher would phone up each participant to ask about any concern or discomfort experienced.
* Monitoring the health parameters such as body temperature, blood pressure, pulse rate, respiratory rate, and urine for routine testing to assess and understand the participants' health condition and detect possible adverse effect of herbal medicines during interim assessment (2nd week of intervention).
* Although very low risk for adverse events (<0.1%), the researcher would terminate the herbal medicine used and ask the participant to attend Accident and Emergency Department immediately if any found such as serious allergy, skin rash or any illness such as fever or systemic infection, which might be related to signs of over reinforcement of Yang inside the body.
* The TCM practitioner will also monitor any uncommon effects on renal and liver functions such as diarrhea, urinary tract infection, pain, and skin rash in the 2nd and 4th week assessments.

Instruments

* Constitution in Chinese Medicine Questionnaire

  o 60 items of Constitution in Chinese Medicine Questionnaire can assess the participants' body constitution.
* Quality of life and symptom severity

  * The 28-item Rhino-conjunctivitis Quality of Life Questionnaire is adopted to evaluate the participants' level of quality of life; and
  * The same questionnaire is also used for assessing their symptoms severity.
* Objective assessment of nasal symptoms
* Peak Nasal Inspiration Flow Meter will be adopted to monitor the nasal symptom (blockage)
* Demographic and other clinical information Pilot Study
* Fifteen participants (i.e. five nursing students in each of three study groups) would be recruited for a pilot study. The pilot study is conducted with the same procedure of TCM assessment, and herbal medicines used.
* Data collection with all the questionnaires, health assessment, follow-ups and data analysis will be performed similar to the main study.
* Purposes of the pilot study are to test the feasibility and procedure of the study, evaluate the validity and reliability of the questionnaires, examine any possible difficulty in sample recruitment and data collection, as well as check the estimated sample size used in the main study. Very minor amendments or modifications have been made on the procedure of the main study according to its results.

Data Collection

* Data collection would be performed at four time points: baseline measurement (Time 1) at recruitment and three post-tests (Times 2-4) (immediately, and 1-month and 3-month following the interventions).
* Baseline assessment would be done to determine the eligibility for participant enrolment (making diagnosis of AR and differentiating their body constitution) and performing baseline measurements (mainly symptom severity, quality of life and body constitution) for the study. After 2-week interim assessment and 4-week intervention, subsequent three post-tests would be performed using the same sets of questionnaires for evaluation of treatment effect and comparison between and within groups.
* All assessments and data collection procedures would be performed in the Integrated Health Clinic, the participants will self-administer the study questionnaires, be assessed by the same TCM practitioner on body constitution and perform other health assessments such as vital signs and urine testing.

ELIGIBILITY:
Inclusion Criteria of the participants are:

1. Nursing students in a full-time bachelor degree program in School of Nursing at The University under study;
2. They are diagnosed by Western medicine and/or TCM practitioner with allergic rhinitis, including those seasonal or perennial one for at least two years;
3. They have a body constitution of Cold and Yang-Deficiency, according to the TCM assessment;
4. They are aged 18 or above and able to speak Cantonese and/or Mandarin; and
5. They can understand written Chinese language, particularly the questionnaires used.

Exclusion Criteria of these students include those who have:

1. A body constitution pattern of Hot and/or Yin-Deficiency, according to the TCM assessment;
2. Currently been taking long-term medications such as anti-hypertensive and psychiatric drugs;
3. Known medical history of co-morbidity of a recent acute and/or chronic disease such as heart, liver and lung disease, cancer, and/or mental illness;
4. Recently undergone major operation(s), are receiving chemotherapy and radiotherapy, or are going to be admitted into hospital over the study period; and
5. Known allergy history of Chinese herbal medicine .

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 298 (Actual)
Dates: Start 2012-06; Primary Completion 2014-08 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Rhino-conjunctivitis Questionnaire (symptom severity) | Baseline
  10cm visual analogue scale used in a 28-item questionnaire to evaluate their symptoms severity.
Rhino-conjunctivitis Questionnaire (symptom severity) | Immediately after intervention (1-2 min)
  10cm visual analogue scale used in a 28-item questionnaire to evaluate their symptoms severity.
Rhino-conjunctivitis Questionnaire (symptom severity) | 1 month after intervention
  10cm visual analogue scale used in a 28-item questionnaire to evaluate their symptoms severity.
Rhino-conjunctivitis Questionnaire (symptom severity) | 3 months after intervention
  10cm visual analogue scale used in a 28-item questionnaire to evaluate their symptoms severity.

SECONDARY OUTCOMES:
Rhino-conjunctivitis Quality of Life Questionnaire | Baseline
  A 28-item health-related-quality of life questionnaire will be used to evaluate QOL.
Constitution in Chinese Medicine Questionnaire | Baseline
  A 60-item questionnaire assesses the participants' patterns of body constitution.
Rhino-conjunctivitis Quality of Life Questionnaire | Immediately after intervention (1-2 min)
  A 28-item health-related quality of life questionnaire will be used to evaluate the participants' disease-specific quality of life.
Rhino-conjunctivitis Quality of Life Questionnaire | 1 month after intervention
  A 28-item health-related quality of life questionnaire will be used to evaluate the participants' disease-specific quality of life.
Rhino-conjunctivitis Quality of Life Questionnaire | 3 months after intervention
  A 28-item health-related quality of life questionnaire will be used to evaluate the participants' disease-specific quality of life.
Constitution in Chinese Medicine Questionnaire | Immediately after intervention (1-2 min)
  A 60-item questionnaire will be used to assess the participants' patterns of body constitution.
Constitution in Chinese Medicine Questionnaire | 1 month after intervention
  A 60-item questionnaire will be used to assess the participants' patterns of body constitution.
Constitution in Chinese Medicine Questionnaire | 3 month after intervention
  A 60-item questionnaire will be used to assess the participants' patterns of body constitution.

OTHER OUTCOMES:
Health assessment | Baseline
  Basic vital signs, urine test, and respiratory functions
Health assessment | Immediately after intervention (1-2-min)
  Basic vital signs, urine test, and respiratory functions will be taken.
Health assessment | 1 month after intervention
  Basic vital signs, urine test, and respiratory functions will be taken.
Health assessment | 3 months after intervention
  Basic vital signs, urine test, and respiratory functions will be taken.

CONTACTS AND LOCATIONS:
Overall Officials: Wai Tong Chien, Principal Investigator — Professor
Locations (1):
- School of Nursing, The Hong Kong Polytechnic University, Hung Hom, Kowloon, Hong Kong

REFERENCES:
- [Background] Jung JW, Kang HR, Ji GE, Park MS, Song WJ, Kim MH, Kwon JW, Kim TW, Park HW, Cho SH, Min KU. Therapeutic effects of fermented red ginseng in allergic rhinitis: a randomized, double-blind, placebo-controlled study. Allergy Asthma Immunol Res. 2011 Apr;3(2):103-10. doi: 10.4168/aair.2011.3.2.103. Epub 2011 Feb 14. PMID 21461249
- [Background] Yang SH, Yu CL, Chen YL, Chiao SL, Chen ML. Traditional Chinese medicine, Xin-yi-san, reduces nasal symptoms of patients with perennial allergic rhinitis by its diverse immunomodulatory effects. Int Immunopharmacol. 2010 Aug;10(8):951-8. doi: 10.1016/j.intimp.2010.05.008. Epub 2010 May 28. PMID 20546945
- [Result] Chan, R.Y.P., & Chien, W.T. (2013). Concepts of body constitution, health and sub-health from traditional Chinese medicine perspective. World Journal of Translational Medicine, 2(3), 56-66. (doi:10.5528/wjtm.v2.i3.56).
- [Result] Chan RY, Chien WT. The effects of two Chinese herbal medicinal formulae vs. placebo controls for treatment of allergic rhinitis: a randomised controlled trial. Trials. 2014 Jul 2;15:261. doi: 10.1186/1745-6215-15-261. PMID 24986270